CLINICAL TRIAL: NCT01916174
Title: A Trial to Demonstrate Bioequivalence Between Two Insulin Degludec/Liraglutide Formulations, B5 and V2 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN9068-4026; 2012-005468-93 (EudraCT Number); U1111-1137-3809 (Other: WHO)
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin degludec/liraglutide, B5 (Experimental): Subjects will be randomly allocated to the two single dose administrations (one for each of the two IDegLira formulations) on the two separate dosing visits. The two administration days will be separated by a wash-out period of 7-15 days.
  Interventions: Drug: insulin degludec/liraglutide
- Insulin degludec/liraglutide, V2 (Experimental): Subjects will be randomly allocated to the two single dose administrations (one for each of the two IDegLira formulations) on the two separate dosing visits. The two administration days will be separated by a wash-out period of 7-15 days.
  Interventions: Drug: insulin degludec/liraglutide

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Subject will receive a single injection (s.c.) of IDegLira B5
  Arms: Insulin degludec/liraglutide, B5
Drug: insulin degludec/liraglutide — Subject will receive a single injection (s.c.) of IDegLira V2
  Arms: Insulin degludec/liraglutide, V2

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess the expected biological equivalence between two formulations of insulin degludec/liraglutide (IDegLira) with identical active ingredient in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers
* Body mass index (BMI) between 18.5 and 27.0 kg/m^2 (both inclusive)
* Body weight between 60 and 90 kg (both inclusive)

Exclusion Criteria:

* Female of child-bearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods. Adequate contraceptive measures are implants, injectables, combined oral contraceptives, hormonal intrauterine device, sexual abstinence or vasectomised partner
* History or presence of cancer, or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrine (incl. diabetes), haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders
* Use of any prescription or non-prescription medication, except for paracetamol, acetylsalicylic acid, contraceptives and vitamins (but including mega-dose vitamin therapy, as judged by the investigator) within 2 weeks before the trial
* Drug or alcohol abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Area under the serum IDeg concentration time curve after single dose | Assessed from 0 to 120 hours
Maximum observed serum IDeg concentration after single dose | Assessed from 0-120 hours
Area under the plasma liraglutide concentration time curve after single dose | Assessed from 0-72 hours
Maximum observed plasma liraglutide concentration after single dose | Assessed from 0-72 hours

SECONDARY OUTCOMES:
Area under the serum IDeg concentration time curve after single dose | Assessed from 0-120 hours
Time to maximum IDeg concentration | Assessed from 0-120 hours
Terminal elimination half-life for IDeg after single dose | Assessed from 0-120 hours
Area under the plasma liraglutide concentration time curve after single dose | Assessed from 0-72 hours
Time to maximum plasma liraglutide concentration after single dose | Assessed from 0-72 hours
Terminal elimination half-life of liraglutide after single dose | Assessed from 0-72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com